CLINICAL TRIAL: NCT02032199
Title: A Prospective Analysis of Changes in Health-Related Quality of Life Following Roux-en-Y Gastric Bypass.
Brief Title: Quality of Life Following Gastric Bypass Surgery.
Status: Completed | Type: Observational
Sponsor: René Klinkby Støving (Other)
Responsible Party: Sponsor-Investigator, René Klinkby Støving, MD, PhD, associate professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: nbhsf36
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: Gastric bypass; Health-related quality of life; SF-36; Questionnaire; Treatment guidelines
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A central goal of health care is to maximize patient functioning and well-being. This has prompted measurement of health-related quality of life (HRQOL) that encompasses physical, psychological, and social functioning. While obese people have generally impaired HRQOL, people seeking bariatric surgery for obesity appear to have poorer HRQOL than obese individuals seeking non-surgical treatment or obese individuals not seeking weight-loss treatment. HRQOL improves significantly after bariatric surgery, but often with large individual variations in outcome. As gastric bypass is an invasive procedure with irreversible influences on eating behaviour and possible serious adverse events, it is important to identify potential risk factors for a poorer long-term result. In Denmark, bariatric surgery is free of charge for patients fulfilling the Danish Health and Medicines Authority guidelines, which until 2011 were in line with international guidelines. However, in 2011 access to surgery was dramatically restricted and the annual number of operations reduced from 0.9 per 1000 inhabitants (2010) to 0.2 per 1000 inhabitants (2012). The restrictions involved a tightening of the criteria for patients without manifest obesity comorbidities, raising lower body mass index (BMI) threshold from 40 to 50 and increasing the lower age limit from 18 to 25 years (11). It is not known whether patients fulfilling the tighter criteria benefit more from surgery than patients who only met the previous criteria.

This study assessed HRQOL changes associated with Roux-en-Y gastric bypass with follow-up over an average of 22 months. The aim was to explore whether postoperative HRQOL variations were associated with identifiable socio-demographic or clinical characteristics. In particular, whether HRQOL changes differed for patients fulfilling the current Danish criteria and patients only fulfilling the previous criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for gastric bypass.

Exclusion Criteria:

* Patients who did not fulfill the national criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients treated with Roux -en-Y gastric bypass surgery in 2008-2010 i Region of Southern Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
36-Item Short Form Health Survey v2 (SF-36) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, PhD, Principal Investigator — Odense Univesity Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Hansen NB, Gudex C, Stoving RK. Improvement in health-related quality of life following Roux-en-Y gastric bypass. Dan Med J. 2014 Jul;61(7):A4870. PMID 25123120